CLINICAL TRIAL: NCT06581913
Title: Investigation of Eating Awareness, Acceptance of Eating Cravings, Wellness Awareness and Health Perception in Healthy Young Adults
Brief Title: Investigation of Eating Awareness,Eating Cravings, Wellness Awareness and Health Perception
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Asli Demirtaş, Lecturer, Nigde Omer Halisdemir University
Other Study IDs: 2024/07-58
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy Young Adults
Keywords: students; awareness; eating; perception
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy young people: Healthy young people aged 18-30 years
  Interventions: Other: Behavioral assessment

INTERVENTIONS:
Other: Behavioral assessment — Eating Awareness, Acceptance of Food Cravings, Healthy Life Awareness Health Perception

SUMMARY:
In this project, eating awareness, acceptance of food cravings, healthy life awareness and health perception will be examined in healthy young adults.

DETAILED DESCRIPTION:
In this project, eating awareness, acceptance of eating desire, healthy life awareness and health perception will be examined in healthy young adults. Accordingly, 356 healthy young individuals between the ages of 18-30 will be included in the study. The questionnaires and scales used as data collection tools in this research, which is planned as a survey study, will be filled in by face-to-face interview method after the written and verbal voluntary consent of the individuals is obtained. The evaluation consists of five sections. It is aimed to raise awareness about the conditions that are found to be related.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old

Exclusion Criteria:

* Under 18 years old
* not volunteering

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young individuals
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Eating Awareness, | Baseline
  Eating Awareness Scale (EAS-30): There are 28 questions, 4-point Likert scale and 5 sub-factors. The Turkish version of the Eating Awareness Scale was used. In the new adapted scale, a 5-point Likert scale was used (1: never, 2: rarely, 3: sometimes, 4: often, 5: always). The high score obtained from each sub-factor of the scale indicates that the individual has the characteristic evaluated by that sub-factor.
Acceptance of Food Cravings, | Baseline
  The Food Craving Acceptance and Action Questionnaire (FAAQ): designed to assess individuals' food craving and food acceptance. The scale is a 6-point Likert-type, 10-item scale. The total score to be obtained from the scale is in the range of 10-60.
Healthy Life Awareness | Baseline
  Health Life Awareness Scale (HLAS) consists of 15 statements and 4 dimensions. The lowest score to be taken from the scale is 15 and the highest score is 75. A high score from the scale is considered as a high level of healthy life awareness. Healthy Life Awareness Scale is a 5-point Likert-type scale. The answers given by the participants are 1: Strongly disagree, 2: Disagree, 3: Undecided, 4: Agree and 5: Strongly Agree and 5: Strongly Agree.
Health Perception | Baseline
  Health Perception Scale (HPS): It is a five-point Likert-type scale consisting of 15 items and four sub-factors. The minimum score that can be obtained from the scale is 15 and the maximum score is 75.
descriptive assessment | Baseline
  In the general information form of the young individuals participating in the study, demographic information (gender, age, height, body weight, body mass index, etc.) was included.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gökçe İnbaşı, MSc., Principal Investigator — Nigde Omer Halisdemir University
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Bor, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study data will not be shared with third parties. The informed consent form has been prepared and approved in this way.